CLINICAL TRIAL: NCT01372618
Title: Breast Cancer Chemoprevention by SOM230, an IGF-I Action Inhibitor
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI has passed away. Requested by department to terminate study.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-00641; BC097854 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2011-06-09; First posted 2011-06-14 (Estimated); Results first posted 2017-12-27 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-11

CONDITIONS: Ductal Carcinoma in Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOM 230/Pasireotide (Experimental): Treatment with SOM230 600mcg twice daily for 20 days.
  Interventions: Drug: SOM 230 / Pasireotide

INTERVENTIONS:
Drug: SOM 230 / Pasireotide — SOM230/Pasireotide is a multi-receptor targeted somatostatin analogue. In this trial, 600 mcg of SOM230/Pasireotide are taken twice daily subcutaneously.

SUMMARY:
This will be a proof of principle clinical trial to evaluate the use of pasireotide (SOM230) in women with ductal carcinoma in situ (DCIS) of the breast. Surgery and radiotherapy are used as treatment for DCIS and subsequent treatment with antiestrogens has been effective in reducing the occurrence of invasive breast cancer. Unfortunately, treatment with antiestrogens carries potential serious side effects and toxicities that are intolerable to some patients. Preliminary data suggest that inhibition of IGF-1 action in the breast will be at least as effective as tamoxifen. Pasireotide is a somatostatin analog that prevents mammary development by inhibiting IGF-1 action directly in the mammary gland and also indirectly without causing menopausal symptoms. This study is an expansion of work that we have previously done in women with atypical hyperplasia of the breast, which showed that treatment with pasireotide for 10 days caused a reduction in the cellularity of these precancerous lesions. In our present study, women with DCIS will be treated with pasireotide for 20 days prior to surgical excision. Endpoints will be as follows:

1. To determine whether pasireotide will inhibit cell proliferation and angiogenesis (signs of tumor growth), and stimulate apoptosis (cell death) in surgically excised tissue in comparison to core biopsies from women with estrogen receptor (ER) positive DCIS. Both the core biopsy and surgical excision are standard of care procedures that women with DCIS have regardless of participation in this trial.
2. To use dynamic contrast enhanced MRI to assess patients before and after treatment with pasireotide and evaluate for changes in tumor volume and other tumor related features
3. In our previous study we found that many women experienced a slight elevation in blood sugar with 10 days of treatment with pasireotide. Other work has shown that this effect often resolves with greater duration of treatment. We are therefore expanding the duration of treatment in this study to 20 days to assess if the initial hyperglycemia seen with pasireotide improves as treatment duration progresses.

DETAILED DESCRIPTION:
Ductal carcinoma in situ (DCIS) is a direct precursor of invasive breast cancer and is also a marker of an increased chance of developing invasive cancer in the ipsilateral and contralateral breast. Surgery and radiotherapy are used as treatment for DCIS and subsequent treatment with antiestrogens has been effective in reducing the occurrence of invasive breast cancer in DCIS patients. Unfortunately, treatment with antiestrogens carries potential side effects and toxicities. The investigators have data to suggest that inhibition of IGF-I action in the breast will be more effective than antiestrogens, raising hopes it might be effective enough to stand alone as a treatment. Pasireotide is a somatostatin analog that prevents mammary development by inhibiting IGF-I action directly in the mammary gland and also indirectly, without causing menopausal symptoms and signs. As both estrogen (E2) and progesterone (P) require IGF-I in order to act, part of the inhibitory effect of pasireotide is on prevention of estrogen action. The investigators have data that indicate that IGF-I also has direct actions on the breast that are independent of steroid hormones. One example is that IGF-I has a direct stimulatory effect on mammary development in the absence of E2. Additionally, IGF-I has effects on ER-negative tumor cell lines that can be reversed by IGF-I inhibition. If pasireotide inhibited both E2 related and E2 unrelated effects of IGF-I it would likely be more effective than antiestrogens. Preliminary data in rats show that pasireotide, at minimum, can entirely substitute for tamoxifen. To determine whether pasireotide had activities in women at high risk for breast cancer, similar to those observed in rats, the investigators were awarded a DOD Synergistic Idea grant. Those data are expected to be reported soon.

The investigators plan to expand this work to determine in principle whether pasireotide has the potential to treat DCIS. The investigators plan on treating 24 women, with low grade (8), intermediate grade (8) and high grade (8) ER-positive DCIS tumors. The investigators will assess its effect on apoptosis, cell proliferation, angiogenesis, ER and PR and phosphorylation of IGF-IR and IRS-1 before and after 20 days of treatment with pasireotide in core biopsy vs. surgical excision specimens. These endpoints will be measured by specific immunohistochemistry. Simultaneously, the investigators will determine whether IGF-I inhibition will reduce angiogenesis in DCIS using dynamic contrast enhanced MRI (DCE-MRI) at 3.0 Tesla, in addition to mammography. This MRI technique is able to detect early changes of neo-angiogenesis associated with invasive breast cancers and DCIS. Pasireotide should theoretically inhibit angiogenesis in these women, as it does in mice. The DCE-MRI may also show changes in tumor volume, morphologic and kinetic features. Imaging will serve as an additional measure to monitor response to treatment. Results will be correlated with pathology and immunohistochemical endpoints.

In our previous work the investigators noted that there was an increase in blood glucose early after starting pasireotide, but the work of others has indicated that this side effect lasts only several weeks. The investigators found that suppressed levels of insulin (due to pasireotide effect on β cells) began to rise by day 10 of treatment. Therefore, extending the treatment period from 10 to 20 days with daily monitoring of patients will enable us to make certain that the early elevated glucose associated with pasireotide is only temporary. Another side effect is reduction in circulating levels of IGF-I. Theoretically, this could lead to body changes associated with growth hormone deficiency (GHD). Although, tamoxifen and raloxifene also lower serum IGF-I, and women taking it do not usually complain of symptoms of GHD, this is an issue that must be further investigated. However, if pasireotide is found to be effective in the treatment of DCIS, the benefit would likely outweigh the risk.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and older
* Must sign informed consent, witnessed, and dated prior to entry
* The participant has breast biopsy consistent with Ductal Carcinoma in situ (DCIS)
* Performance Status: ECOG 0-1 unless mobility is limited from chronic physical handicap
* No clinical evidence of other malignancies (except Basal Cell carcinoma)
* Complete blood count, differential and platelet count must be WNL or verified by the study chair to be related to conditions not interfering with normal health status
* Adequate hepatic and renal function (these must be WNL or verified by study chair to be related to conditions not interfering with normal health status)
* Normal fasting glucose
* No history of diabetes
* Medically and Psychologically able to comply with all study requirements
* Accessible for Follow up

Exclusion Criteria:

* Less than 21 years of age
* Known invasive breast cancer of any type
* Bilateral prophylactic mastectomy
* Prior malignancy of any type that occurred less than 5 years previously, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Existing non-malignant disease that would preclude the administration of pasireotide
* Pregnancy: All subjects will have a beta-hCG serum pregnancy test to rule out pregnancy, a history will also be taken to make certain that recent sexual exposure does not put them at risk for pregnancy. If so a second serum pregnancy test will be done. Volunteers will be asked to use barrier contraception during study.
* Tamoxifen or other preventive measures within 6 months
* Serious Psychiatric condition or addictive disorder
* Diabetes or elevated fasting blood sugar either by history or by HgbA1c greater than 6.5% or fasting serum glucose greater than 100mg/dL on screening labs. If fasting serum glucose is greater than 100mg/dL on screening labs, this test will be repeated to confirm the results
* Inability to inject medication or test for finger stick glucose
* Gall bladder disease
* History of cholecystitis without cholecystectomy
* Electrolyte abnormalities (particularly hypokalemia or hypomagnesemia)
* Contraindication for MRI
* If tumor size is < 1cm on mammography and all calcifications are removed on core biopsy the patient will be excluded.

QT related exclusion criteria

* QTcF at screening > 450 msec.
* History of syncope or family history of idiopathic sudden death.
* Sustained or clinically significant cardiac arrhythmias.
* Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block.
* Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
* Concomitant medication(s) known to increase the QT interval.

Hepatic Related Exclusion Criteria

* Baseline Alanine transaminase (ALT) or Aspartate transaminase (AST) > 2x upper limit of normal (ULN) without known complications of metastatic liver disease or primary hepatic disease (e.g. Cushing's disease and Acromegaly studies).
* Baseline Total Bilirubin > 1.5x ULN

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Kleinberg, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOM 230/Pasireotide
Started | 9
Completed | 0
Not Completed | 9
Not completed — PI Died. Study Terminated | 9

BASELINE CHARACTERISTICS:
Population: Study Terminated. No Data analyzed
Arm/Group | SOM 230/Pasireotide
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Cell Proliferation and Apoptosis
Description: Tissue from initial diagnostic breast biopsies will be compared to the remaining tissue excised after treatment with SOM230. Tissue will be stained to measure cell proliferation and apoptosis (cell death).
Time Frame: Before and after 20 days of treatment
Population: PI death. Study terminated
Arm/Group | SOM 230/Pasireotide
Number analyzed (Participants) | 0

2. Secondary Outcome: Effect of SOM 230 / Pasireotide on Tumor Volume and Tumor Kinetics
Description: To determine whether pasireotide prevents angiogenesis in DCIS as it does in the rat mammary gland, we will immunostain tissue samples for Factor VIII to identify vessels in DCIS before and after treatment. Further, using dynamic contrast enhanced MRI (DCE-MRI) we plan to detect changes in angiogenesis in vivo, non-invasively, and also detect effects of pasireotide which theoretically should inhibit vascularity. We propose to evaluate changes in the size of the lesion, changes in the morphologic appearance and kinetic features of the lesion.
Time Frame: Before and after 20 days of treatment
Population: PI death. Study terminated
Arm/Group | SOM 230/Pasireotide
Number analyzed (Participants) | 0

3. Secondary Outcome: Hyperglycemia
Description: In our previous study, we found that women had moderately increased blood sugar early after starting SOM230. In other studies in normal individuals this effect disappeared by a week or two. We found some evidence of improvement during administration. However, extending the treatment period from 9.5 to 19.5 days will enable us to make certain that the early elevated sugar associated with SOM230 is only temporary.
Time Frame: Before and after 20 days of treatment with 3 month post-treatment follow-up
Population: PI death. Study terminated
Arm/Group | SOM 230/Pasireotide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | SOM 230/Pasireotide
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes